CLINICAL TRIAL: NCT02815930
Title: Characterizing the Senior High Cost User in Ontario: A Population-Based Matched Cohort Study
Brief Title: Characterizing the Senior High Cost User (HCU) in Ontario
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Ontario Drug Policy Research Network (ODPRN) (Unknown); Research Institute of St. Joseph's Hamilton (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2016 0760 236 000
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2019-03

CONDITIONS: Senior High Cost Users (HCU)
Keywords: High cost user (HCU); Healthcare utilization; Healthcare expenditures; Medication use; Medication expenditures; Multimorbidity; Observational study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- HCUs: Newly incident seniors with annual total healthcare expenditures in the top 5% of Ontarians
  Interventions: Other: HCU Status
- Non-HCUs: Seniors with annual total healthcare expenditures below the top 5% of Ontarians

INTERVENTIONS:
Other: HCU Status — Total healthcare expenditures in the top 5% of Ontarians
  Groups: HCUs

SUMMARY:
High cost users (HCUs) are a small group of patients who use a disproportionate amount of health care resources. This study is a retrospective population-based matched cohort analysis of newly incident senior High Cost Users (HCUs) defined as Ontarians aged 66 years or older in the top 5% of healthcare expenditure users in fiscal year 2013 (FY2013). The study objectives are to characterize and contrast Ontario senior HCUs to non-HCUs based on their demographics, co-morbidities, medication use, health service utilization, healthcare expenditures, medication costs and clinical outcomes, and to determine the relative contribution of medications to senior HCUs expenditures

DETAILED DESCRIPTION:
Senior high cost users (HCUs) with annual healthcare expenditures within the top 5% of Ontarians will be identified using established ICES costing algorithms. This cohort will be matched to a cohort of non-HCUs using a 3:1 matching ratio (non-HCU to HCU) based on age at cohort entry (+/- 1 month), sex and geographic location of residence (based on LHIN) for comparative analysis. Descriptive statistics will be used to describe the study populations and outcomes. Regression analyses will be used to adjust for potential confounders when analyzing healthcare resource utilization and costs as a function of HCU status (e.g. income, type of residence, co-morbidities, rural/urban) and/or when analyzing sub-populations [e.g. chronic obstructive pulmonary disease (COPD), congestive heart failure (CHF)]. Logistic regression will be performed using the patient level data to predict the impact of individual factors on the likelihood of becoming a senior HCU.

ELIGIBILITY:
Inclusion Criteria:

* Ontario residents registered in RPDB between April 1, 2013 - March 31, 2014
* Annual total health care expenditures in FY2013 equal to or greater than financial threshold for the top 5% of all Ontarians

Exclusion Criteria:

* Death on OR prior to index date
* Age > 105
* Annual total health care expenditures in FY2012 fiscal year greater than financial threshold of 5% of all Ontarians in FY2013

Ages: 66 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Newly incident senior high cost users (HCUs) in Ontario
Sampling Method: Non-Probability Sample
Enrollment: 700000 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Total healthcare expenditures per patient | 1 year after index date
Total drug costs per patient | 1 year after index date
Drug cost to total healthcare expenditure ratio | 1 year after index date

SECONDARY OUTCOMES:
All-cause mortality | 1 year after index date
All-cause hospitalization rate | 1 year after index date

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lee, BScPhm, ACPR, MD, FRCPC, Principal Investigator — McMaster University

REFERENCES:
- [Derived] Lee J, Muratov S, Tarride JE, Paterson JM, Thavorn K, Mbuagbaw L, Gomes T, Khuu W, Seow H, Thabane L, Holbrook A. Medication use and its impact on high-cost health care users among older adults: protocol for the population-based matched cohort HiCOSTT study. CMAJ Open. 2021 Jan 11;9(1):E44-E52. doi: 10.9778/cmajo.20190196. Print 2021 Jan-Mar. PMID 33436455